CLINICAL TRIAL: NCT00972868
Title: Use of a Novel Unidirectional Face Mask During Noninvasive Positive Pressure Ventilation (NPPV) in Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: A Novel Unidirectional Face Mask During NPPV in COPD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enrole subjucts.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant Professor of Anesthesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000057
Record Dates: First submitted 2009-08-27; First posted 2009-09-09 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Unidirectional mask; NPPV; COPD; respiratory physiology
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD (Experimental): Thirty adult (> 18 years of age) patients in acute hypercapnic respiratory failure resulting from COPD and requiring Noninvasive Positive Pressure Ventilation (NPPV)
  Interventions: Device: A unidirectional face mask (Modified 'Respironics PerformaTrak' Mask)

INTERVENTIONS:
Device: A unidirectional face mask (Modified 'Respironics PerformaTrak' Mask) — The regular face mask will be replaced with the study mask and patients will receive NPPV via the study mask for 30 min. The study mask insures a unidirectional breathing pattern, in through the nose and out through the mouth or in through the mouth and out through the nose. The sequence of these two breathing patterns with opposite flow direction will be chosen randomly. Each will be applied for 30 min with data collected during and at the end of the period.

SUMMARY:
The purpose of this study is to determine the feasibility, safety and efficacy of a unidirectional breathing mask (breathe in through the nose and out through the mouth or breathe in through the mouth and out through the nose) in COPD patients with breathing difficulties requiring noninvasive positive pressure ventilation (NPPV).

ELIGIBILITY:
Inclusion Criteria:

1. Acute hypercapnic respiratory failure as a result of an acute exacerbation of COPD defined as PaCO2 > 50 mmHg, with or without hypoxia, and a respiratory rate of greater than 25/min with the use of accessory muscles of respiration or abdominal paradox;
2. Requiring NPPV as assessed by the managing care team.

Exclusion Criteria:

1. Patients with facial deformity, heavy beard or moustache which prevents a good seal between the mask and the face;
2. Patients who have claustrophobia and cannot wear the mask;
3. Patients who are hemodynamically unstable;
4. Patients who are disoriented and unable to cooperate with the study procedure;
5. DNI or DNR status or patients in whom intubation is contraindicated;
6. Patients who are currently intubated;
7. Patients who recently (< 6months) had an MI or stroke;
8. Pregnant woman; There will be no exclusion based on gender, race or ethnicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in anatomical dead space and improvement in ventilatory efficiency | 30 minutes

SECONDARY OUTCOMES:
Improvement of ventilation rate, tidal volume, end tidal CO2, arterial pH, PaCO2, and PaO2, SpO2, pulse rate, blood pressure and patient rating of comfort of each ventilatory pattern. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital; Robert Kacmarek, PhD, RRT, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States